CLINICAL TRIAL: NCT01749319
Title: Prevention of Baclofen Withdrawal Syndrome: Two-Way Crossover Study of Oral and Intravenous Baclofen in Healthy Adult Volunteers
Brief Title: Oral and IV Baclofen in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Paralyzed Veterans of America Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTSI 20873
Record Dates: First submitted 2012-12-04; First posted 2012-12-13 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Baclofen Withdrawal Syndrome
Keywords: baclofen, withdrawal, interuption, spasticity, pharmacokinetics, tolerability, intravenous, oral
MeSH Terms: conditions — Muscle Spasticity | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Baclofen (Active Comparator)
  Interventions: Drug: Oral baclofen
- Intervenous baclofen (Experimental): Crossover study that eacg subject is given both oral and intervenous baclofen
  Interventions: Drug: Intervenous baclofen

INTERVENTIONS:
Drug: Oral baclofen — Each subject will receive one dose of oral baclofen and one dose of intravenous baclofen on different study days.
  Arms: Oral Baclofen
Drug: Intervenous baclofen
  Arms: Intervenous baclofen

SUMMARY:
The primary objective of this study is to characterize baclofen pharmacokinetics following oral and intravenous administration in patients who are on chronic oral baclofen therapy. The secondary objective is to determine the safety profile of an IV baclofen formulation.

This study is a randomized crossover study with two treatment arms. All subjects will receive a dose of oral baclofen and a dose of IV baclofen on separate study days. Whether the oral or intravenous form is given on the first study day will be randomized in a 1:1 manner.

The pharmacokinetic and tolerability information gained from this study will support the development of further studies to assess the use of IV baclofen to prevent or treat baclofen withdrawal syndrome.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in the study if all of the following conditions exist:

1. Males and females between the ages of 18-65.
2. Subjects are capable of giving informed consent.
3. Female subjects must be post-menopausal for at least 1 year, or surgically incapable of bearing children, or practicing at least one or more of the following methods of contraception for three months prior to, and during the study: hormonal, intrauterine device (IUD), or barrier method in combination with a spermicide.
4. Subject should be medication free, other than study drug, for 48 hours before through 24 hours after study drug administration. If the need for medication is identified during this time period, it will be discussed with and approved by the PI.

   -

Exclusion Criteria:

Subjects will be excluded from participation in the study if any of the following conditions exist:

1. Women who are pregnant.
2. Women who are breast feeding.
3. Subject has a history of intolerance to IV administration of medication.
4. Subject has a known hypersensitivity to baclofen.
5. Subject has a significant history of cardiac, neurologic, psychiatric, oncologic, endocrine, metabolic, renal or hepatic disease
6. Subject has taken or used any investigational drug or device in the 30 days prior to screening.
7. Subject has taken either prescribed or over the counter medication for 48 hours prior to baclofen administration on either of the study days.
8. Subject reveals clinically significant abnormalities on screening laboratory tests.
9. Subject is a non-English speaker, such that ability to ascertain neurological status would require an interpreter.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
oral bioavailability | 5, 15, 30 minutes, and 1, 2, 4, 6, 8, 10, 12, and 24 hours after administration
  oral bioavailability is the fraction of an administered dose of unchanged drug that reaches the systemic circulation
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 5, 15, 30 min and 1, 2, 4, 6, 8, 10, 12, and 24 hours after administration
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Plasma Decay Half-Life (t1/2) | 5, 15, 30 min and 1, 2, 4, 6, 8, 10, 12, and 24 hours after administration
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Maximum concentration (Cmax) | 5, 15, 30 min and 1, 2, 4, 6, 8, 10, 12, and 24 hours after administration
  The maximum concentration is the maximum baclofen concentration observed
Tmax | 5, 15, 30 min and 1, 2, 4, 6, 8, 10, 12, and 24 hours after administration
  Tmax is the time at which the maximum baclofen concentration was observed

SECONDARY OUTCOMES:
assessment of sedation | up to 12 hours
  Sedation will be measured using the Stanford Sleepiness Scale.
Ataxia | up to 12 hours after infusion
  A rating scale of ataxia will be used:
  0=none, 1=mild, 2=severe
  For those who are ambulatory, this will be assessed by gait. Ratings will be:
  mild-unsteady with tandem gait testing, but able to perform without assistance severe-unable to perform tandem gait testing without assistance. For non-ambulatory subjects, ataxia will be assessed by finger to nose and finger pursuit maneuvers.
Nystagmus | up to 12 hours following drug administration
  Nystagmus will be measured using the following scale. 0=none, 1=mild, 2=severe mild-present on extreme gaze; severe-present on midline gaze
blood pressure | 5 minutes immediately prior to, and during the IV infusion and oral administration, then every 15 minutes for 1 hour, then every hour for 12 hours.
  diastolic and systolic blood pressure will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States